CLINICAL TRIAL: NCT07077512
Title: A Single-arm, Phase II Clinical Study of Relmacabtagene Autoleucel Combined With Sintilimab for Relapsed/Refractory B-cell Lymphoma.
Brief Title: Relmacabtagene Autoleucel Combined With Sintilimab for Relapsed/Refractory B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital of Guangzhou Medical University (Other); Guangzhou Overseas Chinese Hospital,Guangdong (Unknown)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-263-01
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Large B Cell Diffuse Lymphoma; Mantle Cell Lymphoma (MCL); Follicular Lymphoma ( FL)
Keywords: Relmacabtagene Autoleucel; Sintilimab; CD19 Positive; B cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell | interventions — relmacabtagene autoleucel; Therapeutics; sintilimab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Relmacabtagene Autoleucel in combination with Sintilimab (Experimental): Patients with CD19-positive relapsed/refractory B-cell lymphoma will receive Relmacabtagene Autoleucel after lymphodepletion therapy (fludarabine + cyclophosphamide) on Day 1. After Relmacabtagene Autoleucel infusion, sintilimab (200 mg IV) will begin on Day 28, administered every 3 weeks until disease progression or intolerable toxicity, with a maximum duration of 1 year.
  Interventions: Drug: Autoleucel (Relmacabtagene Autoleucel); Drug: Sintilimab (PD-1 inhibitor)

INTERVENTIONS:
Drug: Autoleucel (Relmacabtagene Autoleucel) — Relmacabtagene Autoleucel will be reinfused 2 to 7 days after lymphodepletion (fludarabine + cyclophosphamide).
  Other Names: Chimeric Antigen Receptor T-Cell (CAR-T) Therapy
Drug: Sintilimab (PD-1 inhibitor) — Patients will receive intravenous Sintilimab (200 mg every 3 weeks) starting on Day 28 after reinfusion, continuing until disease progression or intolerable toxicity, with a maximum duration of 1 year.
  Other Names: PD-1 Inhibitor

SUMMARY:
This is a prospective, single-arm, multicenter, phase II clinical trial to evaluate the efficacy and safety of Relmacabtagene Autoleucel in combination with the Sintilimab regimen for the treatment of relapsed/refractory B-cell lymphoma

DETAILED DESCRIPTION:
Relmacabtagene Autoleucel treatment: Patients will receive intravenous fludarabine (25 mg/m²/day for 3 days) and cyclophosphamide (250 mg/m²/day for 3 days) for lymphodepletion, with adjustments based on hematologic and renal function.Relmacabtagene Autoleucel will be reinfused 2 to 7 days after lymphodepletion.

Sintilimab treatment: Patients will receive intravenous Sintilimab (200 mg every 3 weeks) starting on Day 28 after reinfusion, continuing until disease progression or intolerable toxicity, with a maximum duration of 1 year.

Primary endpoint: The complete response rate (CRR) at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be aware of and voluntarily sign the informed consent form (ICF).
2. Aged between 18 and 70 years, both male and female.
3. Pathologically diagnosed with DLBCL, FL, or MCL, with histological confirmation of CD19 positivity (immunohistochemistry or flow cytometry, with flow cytometry used for re-evaluation if immunohistochemistry is CD19-negative).
4. The patient must be willing to receive regorafenib and sintilimab treatment and be deemed suitable for this treatment by the investigator.
5. Relapsed/refractory DLBCL, FL, or MCL.
6. At least one measurable or evaluable lesion.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
8. Expected survival of ≥3 months.
9. Adequate function of the heart, lungs, liver, kidneys, and other organs.

Exclusion Criteria:

1. History of another malignancy that has not been in complete remission for at least 2 years, except for: non-melanoma skin cancer, completely resected stage I tumors with low recurrence potential, treated localized prostate cancer, biopsy-confirmed cervical carcinoma in situ, or squamous intraepithelial lesions detected by Pap smear and so on.
2. Active Hepatitis B: a) Positive for Hepatitis B surface antigen (HBsAg) and/or Hepatitis B core antibody (HBcAb) , with HBV-DNA below the lower limit of the reference value can be included.
3. Hepatitis C, HIV, or syphilis infection.
4. Uncontrolled systemic fungal, bacterial, viral, or other infections.
5. Acute or chronic graft-versus-host disease (GVHD).
6. Known hypersensitivity or allergy to any study drug or excipient.
7. Clinically significant central nervous system (CNS) disease or symptoms, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychiatric illness.
8. Pregnant or breastfeeding women, and women of childbearing age who do not wish to use contraception.
9. Mentally ill individuals or those unable to provide informed consent.
10. The investigator deems the patient unsuitable for the study due to medical, psychological, familial, social, or geographical reasons or an inability to comply with the study protocol.
11. Previous CAR-T cell therapy or other gene-modified T-cell treatments.
12. Previous CD19-targeted therapy.
13. Previous allogeneic hematopoietic stem cell transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
The complete response rate (CRR) at 3 months | Up to 3 months after Relmacabtagene Autoleucel infusion

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From the date of the first complete response to the date of the first documented progression or death from any cause, whichever came first,assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Progression-free survival (PFS) | From the date of enrollment until the date of the first documented progression or death from any cause,whichever came first,assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Overall survival (OS) | From the date of enrollment until the date of death from any cause, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Number of participants with adverse events (AE) and severe adverse events (SAE) as assessed by CTCAE v5.0 | Through study completion, an average of 2 years
  To identify the incidence of AE and SAE
Objective Response Rate | Up to 1 year after Relmacabtagene Autoleucel infusion
  To investigate the preliminary anti-tumor efficacy

OTHER OUTCOMES:
Investigating Immune Microenvironment, Proteomic, and Metabolomic Changes Associated with Treatment Efficacy Across Different Patient Group | Through study completion, an average of 2 years
  To investigate the immune microenvironment changes, along with proteomic and metabolomic alterations, and correlate these variations with treatment efficacy across different patient groups.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-sen Universitiy Cancer Center, Guangzhou
  - Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Guangzhou overseas Chinese hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: Undecided